CLINICAL TRIAL: NCT00792714
Title: Determination of the Pharmacokinetics of Inhaled Mannitol After Single and Multiple Dosing in Cystic Fibrosis Patients
Brief Title: Pharmacokinetics of Inhaled Mannitol in Cystic Fibrosis Patients
Acronym: DPM-PK-102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Brett Charlton, Pharmaxis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPM-PK-102
Record Dates: First submitted 2008-11-16; First posted 2008-11-18 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mannitol — 400mg twice daily for 7 days

SUMMARY:
The general objective of the study is to estimate the systemic pharmacokinetics of mannitol after single and multiple dosing of IDPM 400 mg to adult and paediatric cystic fibrosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate in this study in accordance with local regulations
* Have a confirmed diagnosis of cystic fibrosis (sweat test and/or genotype)
* Be aged >6 years (6-11 for paediatrics, 12-17 for adolescents and 18 years for adults)
* Have FEV1 > 30 % and < 90% predicted

Exclusion Criteria:

* Be investigators, site personnel directly affiliated with this study, or their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biologically or legally adopted.
* Be considered "terminally ill" or listed for lung transplantation
* Have had a lung transplant
* Be using nebulised hypertonic saline
* Have had a significant episode of haemoptysis (> 60 mL) in the three months prior to enrolment
* Have had a myocardial infarction in the three months prior to enrolment
* Have had a cerebral vascular accident in the three months prior to enrolment
* Have had major ocular surgery in the three months prior to enrolment
* Have had major abdominal, chest or brain surgery in the three months prior to enrolment
* Have a known cerebral, aortic or abdominal aneurysm
* Be breast feeding or pregnant, or plan to become pregnant while in the study
* Be using an unreliable form of contraception (female patients at risk of pregnancy only)
* Be participating in another investigative drug study, parallel to, or within 4 weeks of study entry (except inhaled mannitol)
* Not able to maintain a mannitol free diet from Day -2 until Day 8 of the treatment phase.
* Have a known allergy to mannitol
* Be using beta blockers
* Have uncontrolled hypertension - systolic blood pressure > 190 and / or diastolic blood pressure > 100
* Have a condition or be in a situation which in the Investigator's opinion may put the subject at significant risk, may confound results or may interfere significantly with the patient's participation in the study
* Be MTT positive.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The general objective of the study is to estimate the systemic pharmacokinetics of mannitol after single and multiple dosing of IDPM 400 mg to adult and paediatric cystic fibrosis patients. | 8 days

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (2):
  - Mater Adult Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Melbourne, Victoria
- United Kingdom (2):
  - Sheffield Children's Clinical Foundation, Sheffield
  - Southampton General Hospital, Southampton